CLINICAL TRIAL: NCT02409875
Title: Baby-STOPP: Targeted Obesity Prevention Directed to Overweight Parents With Young Children
Brief Title: The Early Stockholm Obesity Prevention Project in China
Acronym: ES-China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jianduan Zhang, Associate professor, Huazhong University of Science and Technology
Other Study IDs: ES-2010
Record Dates: First submitted 2015-03-27; First posted 2015-04-07 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Pediatric Obesity
Keywords: early intervention; obesity; body weight; body mass index; overnutrition; early promoters, genetic
MeSH Terms: conditions — Pediatric Obesity; Obesity; Body Weight; Overnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Risk groups: For families that both parents have BMI>=24 or at least one of them BMI>=28, then calculated as high-risk group.
  For families that both parents have BMI<24 or one parents with BMI<24 and one with 24<=BMI<28, then grouped as low-risk group.

SUMMARY:
This is a cohort study where families with infants are followed closely for three years. It aims to assess if parental weight status (normal weight vs. overweight/obesity), their physical activity and eating habit will influence their young children's growth and be helpful in childhood obesity reducing.

DETAILED DESCRIPTION:
The aimed 300 families are invited with half parents in high risk group (one of the parents with BMI>=28 or both 28>BMI>=24) and half in low risk group (both parents with BMI<24 or one parent 28>BMI>=24) living in Wuhan City. Maternal and paternal prepregnancy weight and height are recruited through the Children Systematic Health Management System before the child's first birthday. After getting an oral agreement, a later on family visit will be done by trained staffs. The home visit contains anthropometrics measurement, including weight, height, head circumference, abdominal circumference for both parents and children and blood pressure for parents; it also has some questionnaires that have children's condition during the first years, the caring status, parents' characteristic information, the eating, physical activity and sleeping habits for both parents and children, children's seven day 24 hours' sleeping record in the coming week; at the same time, objectively measured physical activity for parents and children will be done for seven days with accelerometers. The annual visit will range 15 days before or after the children's birthday, and this will begin from the children age one and followed up to aged three.

ELIGIBILITY:
Inclusion Criteria:

* a child in the household being 1 year old (±3 months) at the time of recruitment;
* the parents were Wuhan registered residents;
* the child had no chronic health condition affecting growth, physical activity or eating habits.

Exclusion Criteria:

* none.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families living in Wuhan city, having an one year old child, willing to participanted are welcomed to the study. A total of 300 simple size with half high-risk group and half in low-risk group is anticipated.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-02 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Children BMI | 1 year
  With the annually measured children's weight and height, to calculate the BMI
Children BMI | 2 years
  With the annually measured children's weight and height, to calculate the BMI
Children BMI | 3 years
  With the annually measured children's weight and height, to calculate the BMI

SECONDARY OUTCOMES:
Association between children's eating habit, physical activity level, sleeping pattern and children's BMI | 1 to 3 years
  Using the collected data from questionnaires and accelerometer, to assess the association between the children's eating and physical activity habit with their growth

CONTACTS AND LOCATIONS:
Overall Officials: Jianduan Zhang, Zhang, Study Director — Huazhong University of Science and Technology, Tongji Medical College
Locations (1):
- Tongji Medical College, Wuhan, Hubei, China